CLINICAL TRIAL: NCT01541124
Title: Morphine as the First Drug for the Treatment of Cancer Pain
Brief Title: Morphine as First Drug for Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rioko Kimiko Sakata, Pain Clinic Director, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP1133/07
Record Dates: First submitted 2012-01-10; First posted 2012-02-29 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2012-02

CONDITIONS: Chronic Pain
Keywords: cancer pain; analgesia; morphine
MeSH Terms: conditions — Chronic Pain; Cancer Pain; Agnosia | interventions — Analgesics, Opioid; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Morphine, Pain intensity (Experimental): For cancer pain treatment, World Health Organization recomends tritation of opioids associated with non steroidal antiinflamatory drugs. This study compares the analgesic effect with diferents dosages in 63 patients with cancer pain.
  Interventions: Drug: Opioid

INTERVENTIONS:
Drug: Opioid — 10 mg/pill, po, each 6h, during 6m
  Other Names: Morphine

SUMMARY:
Background and Objectives:

The drugs used as recommended by the WHO does not promote pain relief for all patients with cancer pain. The objective of this study was to evaluate the use of morphine as the first drug for the treatment of moderate cancer pain by visual analogue scale in patients with advanced disease and / or metastases, as an alternative to the recommendations of the WHO analgesic ladder advocated. Methods: The patients without opioid therapy with more than 18 years, were randomly divided into two groups. G1 patients received medication according to the analgesic ladder, starting treatment with non-opioid in the first step, the second weak opioid and opioid potent in the third, and G2 received morphine as first analgesic. There was evaluated the efficacy and tolerability of initial use of morphine every 2 weeks for 3 months. Results: The study was performed in 63 patients. The groups had similar demographics.

DETAILED DESCRIPTION:
After approval of the Ethics Committee and signing the consent, a prospective randomized study was performed in patients ≥ 18 years, with locally advanced cancer and / or metastases, and pain intensity ≤ 6. There were excluded patients with difficulty maintaining clinical follow-up, cognitive impairment and prior treatment with opioids. G1 patients were treated according to the guidelines of the WHO analgesic ladder starting at the first step, with paracetamol 1g each 6 hours, maximum dose of 4 g/ day, in the second, codeine (30 mg each 4 hours , maximum dose 360 mg / day and morphine 10 mg each 4 hours in the third step. Patients in G2 started with morphine 10 mg each 4 hours. Adjuvant drugs have been associated when indicated. According to the intensity of pain the medication was changed according to analgesic ladder in G1 patients and adjusted the dose in G2. The cancer therapy as palliative radiotherapy, chemotherapy or hormone therapy was performed by the oncologist.

There were evaluated: pain intensity every 2 wk. by visual analogue scale (VAS), quality of life every 4 wk. through the brief questionnaire of quality of life of the WHO 19, satisfaction with treatment, physical capacity measured by the index of Eastern Cooperative Oncology Group (ECOG) 20, and the need for additional analgesics. Adverse effects were recorded. The study was considered completed with the patient's death or three months of follow-up.

To calculate the minimum sample size was used the program BioEstat 2.0. There were used as reference means and standard deviations values of study with a similar method 5. Considering a confidence level of 95% study power of 80% of the minimum sample of 30 patients for each group, totaling 60 patients. For the statistical analysis was used GraphPad Prism ®. There was used the Student t test for age, weight, height, chi-square test for patient satisfaction, need for complementation, and adverse effects, and Mann-Whitney test for pain intensity, quality of life and physical capacity. A p value of ≤ 0,05 was considered significant. The resultas were expressed as mean ± DP.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years, with locally advanced cancer and / or metastases, and pain intensity ≤ 6

Exclusion Criteria:

* patients with difficulty maintaining clinical follow-up,
* cognitive impairment and prior treatment with opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Analgesic effect | 3 months
  evaluate the use of morphine as the first drug for the treatment of moderate cancer pain by visual analogue scale in patients with advanced disease and / or metastases, as an alternative to the recommendations of the WHO analgesic ladder advocated

CONTACTS AND LOCATIONS:
Overall Officials: Rioko K Sakata, MD, PhD, Principal Investigator — Universidade Federal de São Paulo
Locations (1):
- Universidade Federal de São Paulo, São Paulo, Brazil